CLINICAL TRIAL: NCT00701701
Title: An Exploratory Study of the Safety and Efficacy of Immune Tolerance Induction (ITI) in Patients With Pompe Disease Who Have Previously Received Myozyme
Brief Title: Immune Tolerance Induction Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was conducted to fulfill a post marketing commitment (PMC 6). FDA acknowledged fulfillment of PMC.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC12817; AGLU03707 (Other: Genzyme Corporation); 2015-000583-34 (EudraCT Number)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II (GSD-II); Glycogenesis 2 Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A: Alglucosidase alfa and Cyclophosphamide (Experimental): Participants exhibiting clinical decline since starting alglucosidase alfa (Myozyme®) therapy and having inhibitory antibodies and/or a sustained high recombinant human acid alpha-glucosidase (rhGAA) antibody titer (defined as at least 2 titers greater than or equal to [>=] 25,600 obtained at least 1 month apart), regardless of their CRIM status, were assigned to Regimen A. In Regimen A, participants received alglucosidase alfa (Myozyme®) Intravenous (IV) infusion of 20 milligram per kilogram (mg/kg) every other week (qow) for a minimum of 18 months or, until the participant reached the age of 2 years (if the participant was less than [<6] months of age at the time of enrollment). In addition, cyclophosphamide 250 milligram per square meter (mg/m^2) IV infusion was administered every 4 weeks (q4w) after Myozyme® infusion for 6 months.
  Interventions: Biological: Myozyme® (alglucosidase alfa)
- Regimen B: Alglucosidase alfa, Rituximab and Methotrexate (Experimental): CRIM-negative participants were assigned to Regimen B if they either(1)exhibited clinical decline since starting alglucosidase alfa (Myozyme®)therapy and did not have inhibitory antibodies and/or a sustained rhGAA antibody titer(defined as at least 2 titers >=25,600 obtained at least 1 month apart),or(2) did not exhibit clinical decline since starting alglucosidase alfa(Myozyme®) therapy, regardless of their anti-rhGAA or inhibitory antibody status. Regimen B participants with CRIM-negative status received alglucosidase alfa(Myozyme®) IV infusion of 20 mg/kg qow for a minimum of 18 months or,until participant reached the age of 2 years (if participant was <6 months of age at time of enrollment). In addition,rituximab 375 mg/m^2 IV was administered weekly beginning the day after Myozyme® infusion for 4 weeks(an optional 2nd cycle could be administered at the discretion of the investigator) and biweekly methotrexate 15 mg/m^2 subcutaneous on the day after Myozyme® infusion for 6 months.
  Interventions: Biological: Myozyme® (alglucosidase alfa)

INTERVENTIONS:
Biological: Myozyme® (alglucosidase alfa) — Myozyme®: IV infusion of 20 mg/kg qow; Cyclophosphamide: 250 mg/m^2 IV q4w after Myozyme infusion for 6 months.
  Other Names: Myozyme®
  Arms: Regimen A: Alglucosidase alfa and Cyclophosphamide
Biological: Myozyme® (alglucosidase alfa) — Myozyme®: IV infusion of 20 mg/kg qow; Rituximab: 375 mg/m^2 IV weekly beginning the day after Myozyme infusion for 4 weeks (an optional additional 2nd cycle could be administered at the discretion of the investigator); Methotrexate: 15 mg/m^2 subcutaneous qow on the day after Myozyme infusion for 6 months.
  Other Names: Myozyme®
  Arms: Regimen B: Alglucosidase alfa, Rituximab and Methotrexate

SUMMARY:
An exploratory, open-labeled study of participants with Pompe disease, who had previously received Myozyme® (alglucosidase alfa) treatment, to evaluate the efficacy, safety and clinical benefit of 2 Immune Tolerance Induction (ITI) regimens in combination with Myozyme®. Eligible participants who were then receiving Myozyme® therapy were enrolled into the study, and were followed for a minimum of 18 months on-study (a 6-month ITI treatment module and a 12-month follow-up module on Myozyme® alone). Eligible participants were followed for a minimum of 18 months on treatment or, if a participant was <6 months of age at the time of enrollment, until the participant was 2 years of age. Both cross-reacting immunologic material (CRIM)-negative and CRIM-positive participants were eligible for Regimen A depending if they met the required criteria. Regimen B, however, was limited to CRIM-negative participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant (and/or participant's legal guardian if participant was < 18 years) provided written informed consent prior to any study-related procedures that were performed.
* The participants had a confirmed diagnosis of Pompe disease defined as a documented acid α-glucosidase (GAA) enzyme deficiency from any tissue source or 2 GAA gene mutations.
* The participant (and/or legal guardian) had ability to comply with clinical protocol.
* If the participant was CRIM-positive, he/she had received at least 6 consecutive months of Myozyme® infusions (20 mg/kg qow).
* If the participant was CRIM-negative, he/she had received at least 1 Myozyme® infusion prior to enrollment.
* Regimen A only: The participants exhibits clinical decline; The participant had persistent high anti-recombinant human acid α-glucosidase (anti-rhGAA) antibody titers and/or tested positive for antibodies that inhibit enzymatic activity and/or uptake of Myozyme®;
* Regimen B only: The participant was CRIM-negative AND The participant did not exhibit clinical decline; OR all of the following: The participant was CRIM-negative AND The participant exhibited clinical decline AND The participant did not exhibit high anti-rhGAA antibody titers and had not tested positive for antibodies that inhibit enzymatic activity and/or uptake of Myozyme®.

Exclusion Criteria:

* The participant had a clinical condition unrelated to Pompe disease that would interfere with program assessments.
* The participant was at risk of reactivation or was a carrier of Hepatitis B or Hepatitis C.
* The participant was at risk of reactivation or had positive serology suggestive of active infection for cytomegalovirus, Herpes simplex, JC virus, Parvovirus or Epstein Barr virus.
* The participant was at risk of reactivation of tuberculosis or had regular contact with individuals who were being actively treated for tuberculosis.
* The participant had low serum albumin.
* The participant had a major congenital abnormality.
* The participant had used any investigational product (other than alglucosidase alfa) within 30 days prior to study enrollment.
* The participant was pregnant or lactating.
* The participant has had or was required to have any live vaccination within one month prior to enrollment.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12-14 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- United States (4):
  - Louisville, Kentucky
  - Durham, North Carolina
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 countries. A total of 5 participants were screened between 14 December 2008 and 17 August 2010 (dates when first participant and last participant signed informed consent), of which one participant died before enrollment.
Pre-assignment Details: A total of 4 participants were included and treated in this study. Participants were assigned to either Regimen A or Regimen B.
Groups:
- Regimen A: Alglucosidase Alfa and Cyclophosphamide: Participants exhibiting clinical decline since starting alglucosidase alfa (Myozyme®) therapy and having inhibitory antibodies and/or a sustained high recombinant human acid alpha-glucosidase (rhGAA) antibody titer (defined as at least 2 titers greater than or equal to [>=] 25,600 obtained at least 1 month apart), regardless of their cross-reacting immunologic material (CRIM) status, were assigned to Regimen A. In Regimen A, participants received alglucosidase alfa (Myozyme®) Intravenous (IV) infusion of 20 milligram per kilogram (mg/kg) every other week (qow) for a minimum of 18 months or, until the participant reached the age of 2 years (if the participant was less than [<6] months of age at the time of enrollment). In addition, cyclophosphamide 250 milligram per square meter (mg/m^2) IV infusion was administered every 4 weeks (q4w) after Myozyme® infusion for 6 months.
Period: Overall Study
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Started | 1 | 3
Completed | 1 | 1
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population is based on full analysis set which included participants who signed informed consent, completed all baseline assessments, and received at least 1 dose of alglucosidase alfa.
Groups:
- Regimen A: Alglucosidase Alfa and Cyclophosphamide: Participants exhibiting clinical decline since starting alglucosidase alfa (Myozyme®) therapy and having inhibitory antibodies and/or a sustained high rhGAA antibody titer (defined as at least 2 titers >=25,600 obtained at least 1 month apart), regardless of their CRIM status, were assigned to Regimen A. In Regimen A, participants received alglucosidase alfa (Myozyme®) IV infusion of 20 mg/kg qow for a minimum of 18 months or, until the participant reached the age of 2 years (if the participant was <6 months of age at the time of enrollment). In addition, cyclophosphamide 250 mg/m^2 IV infusion was administered q4w after Myozyme® infusion for 6 months.
- Total: Total of all reporting groups
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 0 | 2 | 2
  Children (2-11 years) | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was defined as any undesirable physical, psychological, or behavioral effect experienced by participant during his/her participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not product-related. TEAEs were defined as AEs that occurred or worsened during the on-treatment period (time from the start of investigational medicinal product [IMP] administration up to 18 months). Serious AE (SAE) was any AE that resulted in any of the following outcomes: death, was life-threatening, required or prolonged inpatient hospitalization, persistent or significant disability/incapacity; congenital anomaly; or important medical events that may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed above; and/or new invasive ventilator use.
Time Frame: From Baseline up to 18 months
Population: Analysis was performed on safety set population that included participants who received at least 1 dose of alglucosidase alfa in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 1 | 3
Participants
  Any TEAE | 1 | 3
  Any Treatment-emergent SAE | 1 | 3
  Any TEAE leading to withdrawal from study | 0 | 1
  Any TEAE leading to death | 0 | 1

2. Other Pre Specified Outcome: Number of Participants With Anti-Recombinant Human Acid Alpha-glucosidase (Anti-rhGAA) Immunoglobulin G (IgG) Antibodies at Month 18
Time Frame: Month 18
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Groups:
- Regimen A: Alglucosidase Alfa and Cyclophosphamide: Participants exhibiting clinical decline since starting alglucosidase alfa (Myozyme®) therapy and having inhibitory antibodies and/or a sustained high rhGAA antibody titer (defined as at least 2 titers >= 25,600 obtained at least 1 month apart), regardless of their CRIM status, were assigned to Regimen A. In Regimen A, participants received alglucosidase alfa (Myozyme®) IV infusion of 20 mg/kg qow for a minimum of 18 months or, until the participant reached the age of 2 years (if the participant was <6 months of age at the time of enrollment). In addition, cyclophosphamide 250 mg/m^2 IV infusion was administered q4w after Myozyme® infusion for 6 months.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Recombinant Human Acid Alpha-glucosidase (rhGAA) Inhibitory Antibody at Month 18
Description: Participants with positive anti-rhGAA IgG antibody were planned to be assessed for the presence of inhibitory antibodies (inhibition of enzyme activity and inhibition of enzyme uptake). Enzyme-linked immunosorbent assay (ELISA) was used to measure inhibition of rhGAA enzymatic activity in vitro and a cell-based assay was used to measure the inhibition of the uptake of rhGAA in normal fibroblast cells by flow cytometry.
Time Frame: Month 18
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the date of first IMP administration to the date of death due to any cause.
Time Frame: From randomization until death or study cut-off whichever comes earlier (up to 18 months)
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Number of Participants With Ventilator Use
Time Frame: From Baseline up to 18 months
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Left Ventricular Mass (LVM) Z-Score and LVM Index
Description: LVM Z-score and LVM index were assessed by echocardiograms (ECHOs). LVM Z-Score is an indicator of degree of standard deviations from the mean in a normal distribution. The normal range for LVM Z-Score is -2 to 2. Values <-2 or >2 indicate abnormal LVM Z-Score. Values less than 0 (negative values) indicate a smaller LVM than mean and values higher than 0 indicate a larger LVM than the mean. LVM index is an index value derived by normalizing LVM by body surface area. LVM index provides evidence of cardiomyopathy. LVM index values <65 gram per square meter (g/m^2) were considered as normal and LVM index values >=65 g/m^2 were considered as abnormal.
Time Frame: From Baseline up to 18 months
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Gross Motor Disability Assessed by Gross Motor Function Measure-88 (GMFM-88) Score
Description: GMFM-88 is an 88-item measure to detect gross motor function. It consists of 5 categories: lying and rolling; sitting; crawling and kneeling; standing; and walking, running and jumping. Each item is scored on a 4-point Likert scale (0=cannot do; 1=initiates [<10 percent (%) of the task]; 2=partially completes [10% to <100% of the task]; 3=task completion). The score for each dimension is expressed as a percentage of the maximum score for that dimension. Total score is obtained by adding the percentage scores for each dimension and dividing the sum by the total number of dimensions. Total score ranges from 0% to 100%, where higher scores indicate better motor functions. A total score of <7.5% demonstrates gross motor disability.
Time Frame: From Baseline up to 18 months
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Motor Development Status Assessed by Alberta Infantile Motor Scale (AIMS) Score
Description: AIMS is a 58-item reliable and valid measure of motor development for infants at risk for motor delay. It assesses infant movement in 4 positions (subscales): prone (reciprocal crawling); supine (moving hands to feet); sitting (sitting with arm support); and standing (pulls to stand). For each subscale, items are scored as "observed" or "not observed". Items in observed range create a motor window. When scoring, subscale scores are calculated by giving child credit (1 point) for observed items within motor window in addition to being given credit (1 point) for all of the less mature items before motor window. AIMS total score is calculated by summing scores for 58 items and ranges from 0-58, with lower score indicating less mature motor development and higher score indicating more mature motor development.
Time Frame: From Baseline up to 18 months
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Disability Index Assessed by the Pompe Pediatric Evaluation of Disability Inventory (Pompe PEDI) Score
Description: Pompe PEDI is a disease specific version of PEDI which assesses functional capabilities and performance in children with Pompe disease from 2 months through adolescence.It consists of all items of original PEDI (197 functional skill items in 3 domains: self-care; mobility; and social function) and additional items in functional skills, mobility, and self-care domains to reflect clinically relevant functional skills. Each domain consists of 2 subdomains: functional skill performance and caregiver assistance scale. Norm-based scoring was developed for these additional items, and scoring algorithms for PEDI have been adjusted to reflect additional normative data collected for Pompe PEDI. Total score range for each domain (mean of subdomains) and subdomains ranges from 0-100, higher score indicates higher capability.
Time Frame: From Baseline up to 18 months
Population: Data were not summarized for this exploratory outcome measure due to low number of enrollment of participants.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from first IMP administration up to 18 months
Description: Reported AEs and deaths are treatment-emergent adverse events i.e. AEs that developed/worsened and deaths that occurred during the 'on treatment period' (time from first IMP administration until 18 months). Analysis was performed on safety population.
Arm/Group | Regimen A: Alglucosidase Alfa and Cyclophosphamide | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 3/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: Alglucosidase Alfa and Cyclophosphamide (N=1) | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate (N=3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Thrombosis (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac Hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 1 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (4) | 1 (1)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Viral (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Blood Pressure Decreased (Investigations) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Staphylococcus Test Positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: Alglucosidase Alfa and Cyclophosphamide (N=1) | Regimen B: Alglucosidase Alfa, Rituximab and Methotrexate (N=3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (3)
Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Conductive Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Deafness Bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mixed Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Faecaloma (Gastrointestinal disorders) | 1 (2) | 0 (0)
Faeces Hard (Gastrointestinal disorders) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (4) | 1 (1)
Catheter Site Phlebitis (General disorders) | 1 (2) | 0 (0)
Medical Device Complication (General disorders) | 1 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (10) | 2 (10)
Thrombosis In Device (General disorders) | 0 (0) | 1 (1)
Bacterial Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 3 (3)
Otitis Media Acute (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (7)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Feeding Tube Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (3)
Blood Creatine Phosphokinase Mb Increased (Investigations) | 0 (0) | 1 (3)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (2)
Blood Immunoglobulin M Increased (Investigations) | 0 (0) | 1 (1)
Blood Magnesium Decreased (Investigations) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (2)
Body Temperature Increased (Investigations) | 0 (0) | 3 (10)
Heart Rate Increased (Investigations) | 0 (0) | 1 (4)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte Percentage Decreased (Investigations) | 0 (0) | 1 (1)
Muscle Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil Percentage Increased (Investigations) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (3) | 1 (1)
Urine Output Decreased (Investigations) | 0 (0) | 1 (2)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 2 (2)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 1 (1)
Joint Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Clonus (Nervous system disorders) | 0 (0) | 1 (1)
Hypokinesia (Nervous system disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (5) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Red Man Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (6)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to low number of enrollment and exploratory nature of outcome measure, only safety data were summarized and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2009-10-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT00701701/Prot_000.pdf
  • Statistical Analysis Plan (2012-01-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT00701701/SAP_001.pdf